CLINICAL TRIAL: NCT03220321
Title: Pink and White Esthetic Scores of Polymer-infiltrated-ceramic-network and Lithium Disilicate Implant Hybrid Abutment Crowns: Randomized Clinical Trial
Brief Title: Pink and White Esthetic Scores of Polymer-infiltrated-ceramic-network and Lithium Disilicate Implant Hybrid Abutment Crowns
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Nourhan Mohammed Elsaad Elrifaie, Resident, Cairo University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: PES/WES Vita Enamic
Record Dates: First submitted 2017-07-14; First posted 2017-07-18 (Actual); Last update posted 2017-07-18 (Actual); Status verified 2017-07

CONDITIONS: Dental Implants
MeSH Terms: interventions — VITA Enamic; lithia disilicate

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- IPS e.max hybrid abutment crown (Active Comparator)
  Interventions: Other: Lithium disilicate (IPS e.max) hybrid abutment crown
- VITA Enamic hybrid abutment crown (Experimental)
  Interventions: Other: PICN (VITA Enamic) hybrid abutment crown

INTERVENTIONS:
Other: PICN (VITA Enamic) hybrid abutment crown — Hybrid ceramic
  Arms: VITA Enamic hybrid abutment crown
Other: Lithium disilicate (IPS e.max) hybrid abutment crown — Glass ceramic
  Arms: IPS e.max hybrid abutment crown

SUMMARY:
The aim of this study is to evaluate the effect of polymer-infiltrated-ceramic-network hybrid ceramic on pink and white esthetics in comparison with lithium disilicate.

The research hypothesis is that there will be comparable clinical performance results between polymer-infiltrated-ceramic-network and lithium disilicate hybrid abutment crowns.

ELIGIBILITY:
Inclusion Criteria:

* Literate, capable of reading and signing the informed consent document
* Healthy, free from or with controlled systemic disease
* With acceptable oral health to support implant restorations
* With good bone quality and quantity
* Cooperative, accepting follow up and maintenance sessions
* Having single missing tooth in esthetic zone

Exclusion Criteria:

* Under 18 years old
* Illiterate, unable of comprehending or signing the informed consent document
* Unhealthy with uncontrolled systemic disease
* Pregnancy
* With unfavorable oral state that might affect implant procedure and restoration
* Uncooperative, not willing to return for follow up visits

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 18 (Estimated)
Dates: Start 2017-08 (Estimated); Primary Completion 2018-04 (Estimated); Study Completion 2018-04 (Estimated)

PRIMARY OUTCOMES:
Pink Esthetic Score (PES) | 6 months
  Pink esthetics
White Esthetic Score (WES) | 6 months
  White esthetics

IPD SHARING:
Plan to Share IPD: Undecided